CLINICAL TRIAL: NCT02660931
Title: Pediatric Acute Kidney Injury (AKI) Retrospective, Real-Time and Repository Research
Acronym: PAR4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sara Van Driest, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 130558
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Acute Kidney Injury; Renal Injury; Kidney Disease
Keywords: Pediatrics
MeSH Terms: conditions — Acute Kidney Injury; Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- AKI Risk Notification (Experimental): Patients randomized to this arm will be eligible for an acute kidney injury risk notification, if their calculated risk exceeds the threshold during their inpatient encounter.
  Interventions: Other: AKI Risk Notification
- Usual Care (No Intervention): These patients will receive usual clinical care, with no acute kidney injury risk notification.

INTERVENTIONS:
Other: AKI Risk Notification — When a patient's calculated acute kidney injury risk exceeds the threshold value, the electronic medical record will notify the provider of the risk and that appropriate screening (BMP including serum creatinine) may be indicated.
  Arms: AKI Risk Notification

SUMMARY:
This proposal will incorporate statistical models developed by the investigators to predict risk for acute kidney injury into our electronic medical record system, enabling an alert to notify providers of the risk status. Pediatric inpatients will be randomly assigned to be in the intervention group, for whom the notification will be implemented, or in the control group, who will receive usual care (no notification). The investigators believe the notification will increase appropriate screening for acute kidney injury and reduce the severity of acute kidney injury in the intervention group.

DETAILED DESCRIPTION:
This proposal will incorporate a logistic regression models developed by the investigators to predict risk for acute kidney injury in pediatric intensive care unit and pediatric ward patients into the electronic medical record system, enabling personalized decision support. Real-time surveillance using the risk prediction models will identify pediatric inpatients at increased risk for acute kidney injury. When patients exceed the threshold risk for acute kidney injury, the electronic medical record system will notify providers. Patients will be randomly assigned to be in the intervention group, for whom the notification will be implemented, or in the control group, for whom the notification will not display. The risk notification will be assessed for its impact on outcomes including rates of screening for acute kidney injury and the severity of acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* All admissions to the pediatric intensive care unit or pediatric wards at the Monroe Carell Junior Children's Hospital at Vanderbilt

Exclusion Criteria:

* Prior diagnosis of chronic renal disease, including dialysis and transplant
* Admission to the Neonatal Intensive Care Unit during the current admission

Ages: 28 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12108 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Number of Serum Creatinine Tests Ordered | Admission through Discharge (approximately 2 days to 1 week)
  Measure of efficacy of the clinical decision support to lead to increased screening for acute kidney injury.

SECONDARY OUTCOMES:
Length of Stay (days) | Admission through Discharge (approximately 2 days to 1 week)
  Number of days in hospital for admission.
Acute Kidney Injury Severity (as measured by Kidney Disease Improving Global Outcomes [KDIGO] stage 1, 2 or 3) | Admission through Discharge (approximately 2 days to 1 week)
  Worst stage of AKI during hospital stay.
In-hospital Mortality | Admission through Discharge (approximately 2 days to 1 week)
  If any in cohort.
Renal Replacement Therapy (number requiring RRT) | Admission through Discharge (approximately 2 days to 1 week)
  Determined by ICD10 and CPT codes during admission.

CONTACTS AND LOCATIONS:
Overall Officials: Sara L Van Driest, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No